CLINICAL TRIAL: NCT00495456
Title: Cardiovascular Longitudinal Evaluation & Assessment of Risk Study
Brief Title: Cardiovascular Longitudinal Evaluation & Assessment of Risk (CLEAR) Study
Acronym: CLEAR
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Responsible Party: Principal Investigator, Ingrid Hopper, Senior Lecturer, Monash University
Other Study IDs: CGMC 1-07 (CLEAR)
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Cardiovascular Disease
Keywords: cardiovascular; risk; longitudinal; prospective
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The burden of cardiovascular disease (CVD) is considerable, despite many advances in diagnosis, clinical management and drug therapy. The World Health Organization estimates 30% of global deaths are attributable to CVD and whilst mortality rates in developed countries are falling, it remains the largest single cause of death (WHO, 2007). Nineteen out of every 100 deaths in Australia are attributed to CVD, with an annual cost of $1.47 billion (AIHW, 2006).

Assessing the risk of future cardiovascular events is traditionally based on a number of 'risk-factors' determined by observational clinical studies such as the Framingham cohort. Recent evidence however invalidates their use in both the highest and lowest risk groups and raises questions about applying such methods in changing risk-behaviour. A considerable number of new risk markers have surfaced in recent years (including various biomarkers, pulse wave velocity and measures of arterial function). Unfortunately their long-term predictive capacity is largely unknown, particularly when compared with existing risk factors.

The aims of this study are to provide objective longitudinal data for a wide variety of risk markers both in current use and in development. Participants of current on-going clinical studies at will be approached to lengthen their observation period for the purposes of determining long-term clinical outcomes.

Standard clinical observations and data obtained within the participant's enrolled studies will be collated into an electronic database. All existing and future studies must have individual approval from an appropriate ethics committee with signed consent. The baseline studies and follow-up assessments of this cohort will be correlated with cardiovascular events, hospitalizations and mortality. In addition, volunteers can be directed to appropriate clinical studies in CVD, thereby enhancing recruitment, encouraging good quality clinical studies and advancing knowledge of cardiovascular disease prevention.

DETAILED DESCRIPTION:
Design: Longitudinal cohort study

Objectives:

* Establish a database of cardiovascular risk factors
* Correlate with long-term cardiovascular outcomes
* Assign suitable volunteers to appropriate clinical studies

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years of age

Exclusion Criteria:

* Risk assessment would constitute harm to patient
* Informed consent not obtainable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants of current and future cardiovascular trials at the Centre of Clinical Research Excellence, Department of Epidemiology & Preventive Medicine, Monash University, Melbourne.
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2007-08; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
To assess risk factors for cardiovascular disease. | Annually

CONTACTS AND LOCATIONS:
Overall Officials: Dipak Kotecha, MBChB MRCP, Principal Investigator — Monash University; John Varigos, BSc, Principal Investigator — Monash University
Locations (4):
- Australia (4):
  - Box Hill Hospital, Box Hill, Victoria
  - Caulfield General Medical Centre, Caulfield, Victoria
  - The Northern Hospital, Epping, Victoria
  - Alfred Hospital, Melbourne, Victoria

REFERENCES:
- See also: Centre for Clinical Research Excellence in Therapeutics — http://www.ccretherapeutics.org.au/
- See also: Department of Epidemiology & Preventive Medicine, Monash University — http://www.med.monash.edu.au/epidemiology/